CLINICAL TRIAL: NCT01385319
Title: Zotarolimus-eluting Endeavor Sprint Stent in Uncertain DES Candidates (ZEUS) Study
Acronym: ZEUS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Marco Valgimigli (Other)
Responsible Party: Sponsor-Investigator, Marco Valgimigli, Head of the Catheterization laboratory, Università degli Studi di Ferrara
Organization: Università degli Studi di Ferrara (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZEUS-10-II
Record Dates: First submitted 2011-06-24; First posted 2011-06-30 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Coronary Artery Disease
Keywords: Bare metal stent; zotarolimus eluting stent; triple anti-thrombotic therapy; high bleeding riskduration of dual anti-platelet therapy
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bare metal stent (Active Comparator)
  Interventions: Device: Bare metal stent implantation
- Endeavor sprint stent (Experimental)
  Interventions: Device: zotarolimus eluting stent

INTERVENTIONS:
Device: Bare metal stent implantation — After BMS implantation the duration of dual anti-platelet therapy is a function of the clinical presentation and the bleeding risk a given patient as follows:
  Clopidogrel will be given for 1 month after PCI if indication to the procedure is stable coronary artery disease or for at least 6 month if indication to the procedure is ACS, including STEMI or NSTEACS. At discretion of the treating physician, prasugrel or ticagrelor may replace clopidogrel in ACS patients.
  Patients recruited in the study due to high bleeding risk will receive clopidogrel for at least 30 days.
  Patients recruited in the study due to high thrombosis risk will receive clopidogrel monotherapy life long or DAPT for at least 1 month.
  Arms: bare metal stent
Device: zotarolimus eluting stent — After ZES implantation the duration of dual anti-platelet therapy is a function of the clinical presentation and the bleeding risk a given patient (i.e. identical to criteria set out for BMS patients) as follows:
  Clopidogrel will be given for 1 month after PCI if indication to the procedure is stable coronary artery disease or for at least 6 month if indication to the procedure is ACS, including STEMI or NSTEACS. At discretion of the treating physician, prasugrel or ticagrelor may replace clopidogrel in ACS patients.
  Patients recruited in the study due to high bleeding risk will receive clopidogrel for at least 30 days.
  Patients recruited in the study due to high thrombosis risk will receive clopidogrel monotherapy life long or DAPT for at least 1 month.
  Arms: Endeavor sprint stent

SUMMARY:
To prospectively evaluate in a multicenter open label trial whether the use of zotarolimus-eluting ENDEAVOR Stent implantation in patients at low restenosis or at high bleeding or thrombotic risk will decrease the incidence of 12-month major adverse cardiac events (MACE) including overall death, any myocardial infarction (MI) or any target vessel revascularization (TVR).

DETAILED DESCRIPTION:
The aim of this study is to conduct a multicenter, international, randomized trial to test whether the Endeavor stent is superior to BMS in terms of efficacy and safety in

1. Patients with coronary artery disease lesions at low risk of in-stent restenosis;
2. Patients at high risk for bleeding or carrying impossibility to comply with dual anti-platelet treatment at long-term.
3. Patients at high thrombosis risk due to systemic disorders or planned non-cardiac surgery within 12 months

As the use of DES in these two patient/lesion subsets is debated due to lack of evidence, patients fulfilling at least one of these three medical conditions qualify for bare metal stent implantation and physicians may believe DES to be even contra-indicated in such cases. The current protocol has been developed on purpose to address the value of the Endeavor Sprint stent, which differs in many aspects from other FDA approved DES, including fast and complete degree of strut coverage after implantation and quick release of active drug after deployment (~15 days) which may help decreasing the need for prolonged dual antiplatelet treatment down to 1 month as it is currently recommended for bare metal stent implantation.

ELIGIBILITY:
Inclusion Criteria:

A) low restenosis risk based on angiographic findings defined as follows:

----patients will be considered at low restenosis risk if no planned stent lower than 3.0 mm is intended to be implanted in lesions expect left main or vein graft

B) high bleeding risk and/or presence of relative-absolute contraindication to dual anti-platelet treatment beyond 30 days defined as follows:

1. Clinical indication to treatment with oral anticoagulant, including use of warfarin or dabigatran or other oral anticoagulant agents
2. Recent (within previous 12 months) bleeding episode(s) which required medical attention
3. Previous bleeding episode(s) which required hospitalization if the bleeding diathesis has not been completely resolved (i.e. surgical removal of the bleeding source)
4. Age greater than 80
5. Systemic conditions associated to increased bleeding risk (e.g. hematological disorders or any known coagulopathy determining bleeding diathesis, including history of or current thrombocytopenia defined as platelet count <100,000/mm3 (<100 x 109/L).
6. Known Anemia defined as repeatedly documented hemoglobin lower than 10 gr/dl which is not due to an acute and documented blood loss
7. Need for chronic treatment with steroids or NSAID

C) Patients at high thrombosis risk based on the presence of at least one of the following criteria:

1. Allergy/intolerance to aspirin
2. Allergy/intolerance to clopidogrel AND ticlopidine
3. Planned surgery (other than skin) within 12 months of percutaneous coronary intervention (PCI).
4. patient with cancers (other than skin) and life expectancy >1 year
5. Patients with systemic conditions associated with thrombosis diathesis (e.g., hematologic disorders and any known systemic conditions determining a pro-thrombotic state including immunological disorders)

   -

   Exclusion Criteria:
   * Any of the following:

     1. Women who are pregnant. Women of childbearing potential must have a negative pregnancy test (urine or serum HCG) within 7 days prior to randomization; as close to randomization as possible, within 24 hours preferred.
     2. Subjects who are unable to give informed consent and assurance for complete contact through 12 months.
     3. PCI with stenting in the previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1606 (Actual)
Dates: Start 2011-06; Primary Completion 2012-09 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
MACE | 12 months
  Major adverse cardiovascular events including death for any cause, non-fatal myocardial infarction or target vessel revascularisation

SECONDARY OUTCOMES:
Death | 12 months
myocardial infarction | 12 months
TVR | 12 months
  target vessel revascularisation
stent thrombosis | 12 months

CONTACTS AND LOCATIONS:
Locations (16):
- Albert Szent-Györgyi Clinical Center, University of Szeged, Szeged, Hungary
- Italy (13):
  - Ospedale San Donato, Arezzo, AR
  - Ospedali Riuniti di Bergamo, Bergamo, BG
  - Policlinico San Marco, Zingonia, BG
  - Ospedale di Savigliano, Savigliano, CN
  - Istituto Clinico Sant'Ambrogio, Milan, MI
  - Azienda Unita' Sanitaria Locale Di Modena - Ospedale Baggiovara, Modena, MO
  - Azienda Ospedaliero-Universitaria di Parma, Parma, PR
  - Policlinico San Matteo, Pavia, PV
  - Ospedale di Ravenna, Ravenna, RA
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Ospedale Umberto I, Torino, TO
  - Ospedale San Giovanni Bosco, Torino, TO
  - University Hospital of Ferrara, Ferrara
  - Clinica Mediterranea, Naples
- Hospital de Santa Cruz, Carnaxide, Portugal
- University Hospital of Geneva, Geneva, Switzerland

REFERENCES:
- [Derived] Ariotti S, Adamo M, Costa F, Patialiakas A, Briguori C, Thury A, Colangelo S, Campo G, Tebaldi M, Ungi I, Tondi S, Roffi M, Menozzi A, de Cesare N, Garbo R, Meliga E, Testa L, Gabriel HM, Ferlini M, Vranckx P, Valgimigli M; ZEUS Investigators. Is Bare-Metal Stent Implantation Still Justifiable in High Bleeding Risk Patients Undergoing Percutaneous Coronary Intervention?: A Pre-Specified Analysis From the ZEUS Trial. JACC Cardiovasc Interv. 2016 Mar 14;9(5):426-36. doi: 10.1016/j.jcin.2015.11.015. PMID 26965932
- [Derived] Valgimigli M, Patialiakas A, Thury A, McFadden E, Colangelo S, Campo G, Tebaldi M, Ungi I, Tondi S, Roffi M, Menozzi A, de Cesare N, Garbo R, Meliga E, Testa L, Gabriel HM, Airoldi F, Ferlini M, Liistro F, Dellavalle A, Vranckx P, Briguori C; ZEUS Investigators. Zotarolimus-eluting versus bare-metal stents in uncertain drug-eluting stent candidates. J Am Coll Cardiol. 2015 Mar 3;65(8):805-815. doi: 10.1016/j.jacc.2014.11.053. PMID 25720624
- [Derived] Valgimigli M, Patialiakas A, Thury A, Colangelo S, Campo G, Tebaldi M, Ungi I, Tondi S, Roffi M, Menozzi A, de Cesare N, Garbo R, Meliga E, Testa L, Gabriel HM, Airoldi F, Ferlini M, Liistro F, Dellavalle A, Vranckx P, Briguori C. Randomized comparison of Zotarolimus-Eluting Endeavor Sprint versus bare-metal stent implantation in uncertain drug-eluting stent candidates: rationale, design, and characterization of the patient population for the Zotarolimus-eluting Endeavor Sprint stent in uncertain DES candidates study. Am Heart J. 2013 Nov;166(5):831-8. doi: 10.1016/j.ahj.2013.07.033. Epub 2013 Sep 26. PMID 24176438